CLINICAL TRIAL: NCT02898441
Title: Community-based Early Stage Lung Cancer Screening With Low-dose Computed Tomography in China
Brief Title: Early Stage Lung Cancer Screening With Low-dose Computed Tomographic
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Baohui Han, Vice-President, Shanghai Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2013ZYJB0402
Record Dates: First submitted 2016-09-08; First posted 2016-09-13 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: Lung Cancer
Keywords: lung cancer screening; low-dose CT; high-risk population
MeSH Terms: conditions — Lung Neoplasms | interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Screening Arm (Active Comparator): LDCT was performed at baseline + 2 biennial repeated LDCT rounds
  Interventions: Device: Low Dose Computed Tomography
- Passive Arm (No Intervention): Eligible subjects were randomized to follow up in usual care

INTERVENTIONS:
Device: Low Dose Computed Tomography — LDCT were performed in screening arm. The abnormal nodules were defined as noncalcified nodules (NCN) larger than 4 mm.
  Arms: Screening Arm

SUMMARY:
The present study is a randomized controlled trial of LDCT screening for lung cancer versus usual care. 6000 high-risk subjects (age 45-70) were recruited and randomized to the Active arm (Baseline + 2 biennial repeated LDCT screening) or to the Passive arm, followed up in usual care (Baseline + 2 biennial repeated questionnaire inquiries). Follow-up for lung cancer incidence, lung cancer mortality and overall mortality was performed. Blood samples were stored from the Active arm in a Biobank. Management of positive screening test was carried out by a pre-specified protocol.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants were those aged 45-70 years, and with either of the following risk factors:

  1. history of cigarette smoking ≥ 20 pack-years, and, if former smokers, had quit within the previous 15 years;
  2. malignant tumors history in immediate family members;
  3. personal cancer history;
  4. professional exposure to carcinogens;
  5. long term exposure to second-hand smoke;
  6. long term exposure to cooking oil fumes.

Exclusion Criteria:

1. Had a CT scan of chest within last 12 months
2. History of any cancer within 5 years

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6000 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Lung cancer incidence rate | 5 years
  Assess the number of lung cancer incidences after each round of screening in both arms. Compared the stage differences between screening arm and usual care arm.

SECONDARY OUTCOMES:
Lung cancer mortality | 5 years
  Assess lung cancer mortality in both arms within next 5 years after first round of screening.
All-cause mortality | 5 years
  Assess all-cause mortality in both arms within next 5 years after first round of screening.

OTHER OUTCOMES:
Nodule detection rate | One year
  Assess nodule detection rate, and the types and sizes of nodules detected in LDCT screening arm.

CONTACTS AND LOCATIONS:
Overall Officials: Baohui Han, MD, PhD, Principal Investigator — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided